CLINICAL TRIAL: NCT04389463
Title: Patient Outcome of Cardiac Surgery During the COVID-19 Pandemic ; International Cohort Study
Brief Title: Patient Outcome of Cardiac Surgery During the COVID-19 Pandemic
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HEART-19 Study
Record Dates: First submitted 2020-05-14; First posted 2020-05-15 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Patients Undergoing Cardiac or Thoracic Surgery
Keywords: Cardiac surgery; Postoperative outcome; COVID-19; SARS-Cov 2 infection; Postoperative complication
MeSH Terms: conditions — COVID-19; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cardiac or thoracic surgery in COVID-19 positive patients
  Interventions: Other: No intervention
- Cardiac/thoracic surgery in COVID-19 negative patients
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No description

SUMMARY:
This study will describe the recovery process of patients undergoing cardiac surgery during the covid-19 pandemic. This will focus on hemodynamic failure and organ dysfunction after surgery.

Capturing real-world data and sharing international experience will inform the management of this complex group of patients who undergo surgery throughout the COVID-19 pandemic, improving their clinical care.

This investigator-led, non-commercial, non-interventional does not collect any patient identifiable information.

DETAILED DESCRIPTION:
Performing cardiac surgery in the context of SARS-CoV2 infection is potentially at risk of marked post-operative hemodynamic failure (shock) due to the inflammatory reaction generated by the surgery and the extracorporeal circulation associated with the viral infection. In addition, in the absence of infection, 30-50% of patients will experience acute post-operative respiratory failure due to the combined effects of extracorporeal circulation and general anesthesia. The pulmonary tropism of the virus therefore is susceptible to increase in post-operative respiratory impairment.

Thus, the infection is likely to favor the occurrence of post-operative shock but also to aggravate respiratory failure and other post-operative organ failures.

Therefore, the investigators designed an observational study that aims at comparing two groups of patients:

* Cardiac or thoracic surgery patients with a negative Covid-19 PCR pre-operatively and in the 15 following days
* Cardiac or thoracic surgery patients with a positive Covid-19 PCR in the 15 days before surgery

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years) undergoing cardiac or thoracic surgery
* With positive PCR in the 5 days before or after cardiac/thoracic surgery.

Exclusion Criteria:

* Minors

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac or thoracic surgery during the COVID-19 pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2026-05-11 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Highest VIS (Vasoactive-Inotropic Score) in the first 12 hours postoperatively. | 12 hours post-operatively
  The VIS score correlates with mortality after cardiac surgery and reflects the degree of patient hemodynamic failure. This score is calculated as follows:
  ISR = Dobutamine dose in g/kg/min + 100 times the Adrenaline dose in g/kg/min + 100 times the Noradrenaline dose in g/kg/min + 10,000 times the Vasopressin dose in U/kg/min.

SECONDARY OUTCOMES:
Post-operative organ failure | 5 days post-operatively
  Prospective assessment of ICU outcomes until all included patients were discharged from ICU
Post-operative outcome | 28 days post-operatively
  Prospective assessment of ICU outcomes until all included patients.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No